CLINICAL TRIAL: NCT01856803
Title: Anti-thymocyte Globulins for GVHD Prophylaxis After HLA-matched Sibling Stem Cell Transplantation in Patients at 40 Years of Age or More With Hematological Malignancies
Brief Title: Anti-thymocyte Globulins for Graft-versus-host Disease Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, director of peking university institute of hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-08
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Leukemia, GVHD, ATG, Transplantation
MeSH Terms: conditions — Leukemia; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- routine prophylaxis (Active Comparator): In this group, CSA plus MMF and MTX adopted as prevention of GVHD.
  Interventions: Drug: anti thymoglobulin
- ATG prophylaxis (Experimental): In this group,ATG+MMF+CsA+MTX was adopted as prevention of GVHD
  Interventions: Drug: anti thymoglobulin

INTERVENTIONS:
Drug: anti thymoglobulin

SUMMARY:
Age is a risk factor for graft-versus-host disease (GVHD) after human leukocyte antigen (HLA)-matched sibling allogeneic stem cell transplantation (allo-SCT). The incidence of acute GVHD is significantly higher in patients at 40 years of age or more than those at 18 to 39 years of age after allo-SCT. It was found that Anti-thymocyte globulins can be used for prophylaxis of both acute and chronic GVHD after allo-SCT.Prophylaxis of GVHD using ATG in patients at 40 years of age or more in matched sibling allo-SCT settings might significantly decrease the incidence of acute and chronic GVHD and the incidence of late effect after transplantation.

DETAILED DESCRIPTION:
Prophylaxis for GVHD included CSA, MTX and MMF±ATG. In the trial group, CSA was started intravenously on day -1, at the dosage of 3 mg/kg, and switched to oral formulation as soon as the patient was able to take medication after engraftment. The dosage was adjusted to maintain a trough blood level of 200-300ng/ml. MMF was administered orally, 0.25g every 12 hours, from day -1 before transplantation to day 30 after transplantation. The dosage of MTX was 15 mg/m2, administered i.v. on day 1, and 10 mg/m2 on days 3, 6, and 11 after transplantation. ATG (Thymoglobulin 2.5mg/kg per day i.v.) on days -2 through -1. In the control group, CSA was started intravenously on day -1, at the dosage of 3 mg/kg, and switched to oral formulation as soon as the patient was able to take medication after engraftment. The dosage was adjusted to maintain a trough blood level of 200-300ng/ml. MMF was administered orally, 0.25g every 12 hours, from day -1 before transplantation to day 30 after transplantation. The dosage of MTX was 15 mg/m2, administered i.v. on day 1, and 10 mg/m2 on days 3, 6, and 11 after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Standard-risk of recipients with hematological malignancies (including AML-CR1, ALL-CR1, CML-CP, MDS-RA, RARS,RCMD,RAEB-1); age from 40 to 60; having HLA-matched sibling donor; Eastern Cooperative Oncology Group (ECOG)≤1, ejection fraction (EF)≥50%; bilirubin≤35µmol/L; AST, and ALT lower than or equall to two-fold baseline;creatinie≤130µmol/L.

Exclusion Criteria:

* Active, uncontrolled infection; severe allergy to ATG, including shock or laryngeal edema; secondary stem cell transplant recipient; haplidentical recipients; matched unrelated donor recipients; non-myeloablative condioning regimen recipients; EF<50%; bilirubin>35µmol/L; AST, and ALT higher than two-fold baseline; creatinie>130µmol/L.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GVHD, and chronic GVHD | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189
- [Derived] Chang YJ, Wu DP, Lai YR, Liu QF, Sun YQ, Hu J, Hu Y, Zhou JF, Li J, Wang SQ, Li W, Du X, Lin DJ, Ren HY, Chen FP, Li YH, Zhang X, Huang H, Song YP, Jiang M, Hu JD, Liang YM, Wang JB, Xiao Y, Huang XJ. Antithymocyte Globulin for Matched Sibling Donor Transplantation in Patients With Hematologic Malignancies: A Multicenter, Open-Label, Randomized Controlled Study. J Clin Oncol. 2020 Oct 10;38(29):3367-3376. doi: 10.1200/JCO.20.00150. Epub 2020 Jul 10. PMID 32650683